CLINICAL TRIAL: NCT03901521
Title: Autosomal Dominant Polycystic Kidney Disease Somatic Mutation Biorepository
Acronym: ADPKD
Status: Enrolling by invitation | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: The Rogosin Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 1710018665
Record Dates: First submitted 2019-03-13; First posted 2019-04-03 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Dr. Rennert's Molecular Genetic Research laboratory personnel at the Pathology and Laboratory Medicine Department of Weill Cornell Medicine (WCM) will coordinate the process of sample handling with the surgeon.
  This study will be using native kidney tissue from ADPKD subjects received in the Surgical Pathology Laboratory (Starr 10), at the Department of Pathology and Laboratory Medicine. The kidney tissue will be collected on the day of the native nephrectomy, following examination and clearance by the surgical pathologist. Immediately after the ADPKD kidney is removed, it will be collected in the Operating Room (OR) using a sterile container and a co-investigator will deliver the specimen to Surgical Pathology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will analyze the germline and somatic mutations underlying the development of ADPKD in order to better understand the genetic mechanism responsible for the cystic transformation. Once identified, these mutations could help us understand better the mechanism leading to the development of this disease and may explain at least in part the phenotypic variability.

DETAILED DESCRIPTION:
The presentation of ADPKD renal and extrarenal manifestations varies widely, even within families, and has been attributed to numerous genetic factors. One principal explanation came with the discovery that renal cyst lining cells from ADPKD patients undergo secondary somatic mutations, selective loss of the second copy of a respective normal polycystic kidney disease (PKD) gene. These somatic mutations can occur in either polycystic kidney disease 1 (PKD1) or polycystic kidney disease 2 (PKD2). Furthermore, various cysts in the same patient have been reported to harbor different somatic mutations. These findings implicated a cellular recessive mechanism for cyst formation in ADPKD, suggesting the possibility that the observed intra-familial variation in disease phenotype may, at least in part, be explained by variation in mutation type, the timing and number of somatic "second-hit" mutations in individual family members affected with the disease. However, there is currently very little known about the cellular genetic mechanism leading to cysts development and very few studies, addressing this issue.

ELIGIBILITY:
Inclusion Criteria:

* Males or females
* 18 years of age or older
* Confirmed diagnosis of ADPKD
* Undergoing a native nephrectomy
* Willing and able to provide informed consent

Exclusion Criteria:

* Unable or unwilling to provide informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria include patients with a diagnosis of end-stage renal disease caused by ADPKD who are scheduled for native nephrectomy. The clinical indications for native nephrectomy will be determined by the surgeon prior to enrollment of the subject. These patients will be identified during the pre-operative evaluation that occurs prior to the surgery. At the time of this evaluation, subject eligibility will be assessed by a co-investigator and their willingness to participate will be evaluated. Subjects who agree to participate will provide informed consent, and blood samples (30 mL) will be obtained for extraction of nucleic acids, in addition to the routine preoperative blood tests.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The presence of somatic PKD 1/2 gene mutations in cyst epithelial cells | 10 YEARS
  The presence of mutations will be measured by next generation sequencing (NGS) and other tools for mutation analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Priya Velu, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be shared with other investigators. Data will be de-identified.
Supporting Information: Study Protocol
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Tan AY, Blumenfeld J, Michaeel A, Donahue S, Bobb W, Parker T, Levine D, Rennert H. Autosomal dominant polycystic kidney disease caused by somatic and germline mosaicism. Clin Genet. 2015 Apr;87(4):373-7. doi: 10.1111/cge.12383. Epub 2014 Apr 26. PMID 24641620
- [Background] Tan AY, Zhang T, Michaeel A, Blumenfeld J, Liu G, Zhang W, Zhang Z, Zhu Y, Rennert L, Martin C, Xiang J, Salvatore SP, Robinson BD, Kapur S, Donahue S, Bobb WO, Rennert H. Somatic Mutations in Renal Cyst Epithelium in Autosomal Dominant Polycystic Kidney Disease. J Am Soc Nephrol. 2018 Aug;29(8):2139-2156. doi: 10.1681/ASN.2017080878. Epub 2018 Jul 24. PMID 30042192
- [Background] Zhang Z, Bai H, Blumenfeld J, Ramnauth AB, Barash I, Prince M, Tan AY, Michaeel A, Liu G, Chicos I, Rennert L, Giannakopoulos S, Larbi K, Hughes S, Salvatore SP, Robinson BD, Kapur S, Rennert H. Detection of PKD1 and PKD2 Somatic Variants in Autosomal Dominant Polycystic Kidney Cyst Epithelial Cells by Whole-Genome Sequencing. J Am Soc Nephrol. 2021 Dec 1;32(12):3114-3129. doi: 10.1681/ASN.2021050690. Epub 2021 Dec 1. PMID 34716216
- [Result] Zhang W, Tan AY, Blumenfeld J, Liu G, Michaeel A, Zhang T, Robinson BD, Salvatore SP, Kapur S, Donahue S, Bobb WO, Rennert H. Papillary renal cell carcinoma with a somatic mutation in MET in a patient with autosomal dominant polycystic kidney disease. Cancer Genet. 2016 Jan-Feb;209(1-2):11-20. doi: 10.1016/j.cancergen.2015.11.002. Epub 2015 Dec 1. PMID 26718059
- [Result] Zhang W, Stephens CJ, Blumenfeld JD, Behzadi AH, Donahue S, Bobb WO, Newhouse JH, Rennert H, Zhao Y, Prince MR. Relationship of Seminal Megavesicles, Prostate Median Cysts, and Genotype in Autosomal Dominant Polycystic Kidney Disease. J Magn Reson Imaging. 2019 Mar;49(3):894-903. doi: 10.1002/jmri.26289. Epub 2018 Sep 19. PMID 30230107
- [Result] Tan AY, Michaeel A, Liu G, Elemento O, Blumenfeld J, Donahue S, Parker T, Levine D, Rennert H. Molecular diagnosis of autosomal dominant polycystic kidney disease using next-generation sequencing. J Mol Diagn. 2014 Mar;16(2):216-28. doi: 10.1016/j.jmoldx.2013.10.005. Epub 2013 Dec 27. PMID 24374109
- [Result] Ben-Dov IZ, Tan YC, Morozov P, Wilson PD, Rennert H, Blumenfeld JD, Tuschl T. Urine microRNA as potential biomarkers of autosomal dominant polycystic kidney disease progression: description of miRNA profiles at baseline. PLoS One. 2014 Jan 29;9(1):e86856. doi: 10.1371/journal.pone.0086856. eCollection 2014. PMID 24489795